CLINICAL TRIAL: NCT06128252
Title: A Prospective, Multicentre, Double-blind Randomized Controlled Clinical Study of the Efficacy and Safety of Taurine Combined With Serplulimab and Chemotherapy Versus Serplulimab Combined With Chemotherapy for Treatment of Locally Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Clinical Study of Taurine Combined With Neoadjuvant Chemo-Immunotherapy for Treatment of Locally Advanced Gastric Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K202308-01
Record Dates: First submitted 2023-11-02; First posted 2023-11-13 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Gastric Cancer
Keywords: Taurine; neoadjuvant immunotherapy and chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Taurine; XELOX

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, double-blind, randomized controlled clinical study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taurine + Serplulimab + XELOX (Experimental): Taurine + Serplulimab + XELOX chemotherapy regimen
  Interventions: Dietary Supplement: Taurine; Biological: Serplulimab; Drug: XELOX regimen
- Placebo + Serplulimab + XELOX (Active Comparator): Taurine placebo + Serplulimab + XELOX chemotherapy regimen
  Interventions: Biological: Serplulimab; Drug: XELOX regimen; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Taurine — Taurine supplementation in tablets of 1.0 gram of taurine powder. Dosage: 3.0 gram/day. Frequency: 3 time/day.
  Arms: Taurine + Serplulimab + XELOX
Biological: Serplulimab — Serplulimab
Drug: XELOX regimen — Oxaliplatin + capecitabine
Dietary Supplement: Placebo — Taurine placebo in tablets of 1.0 gram of starch powder. Dosage: 3.0 gram/day. Frequency: 3 time/day.
  Arms: Placebo + Serplulimab + XELOX

SUMMARY:
This project aims to evaluate the efficacy and safety of oral taurine supplementation combined with PD-1 inhibitor (serplulimab) and chemotherapy in inducing systemic CD8+ T cell responses and achieving improved gastric cancer patient outcomes than with serplulimab and chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, no gender limitation;
2. Pathologically confirmed gastric or gastroesophageal junction adenocarcinoma with cTNM stage II/III，T≥3, N ≥0, M=0；
3. Expected survival of ≥ 3 months;
4. The tumor specimens were PD-L1 positive (CPS ≥ 1)；
5. There is a measurable lesion with the possibility of radical R0 resection after evaluation by doctors；
6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
7. Patients informed about the purpose and course of the study and provided a written consent to participate.

Exclusion Criteria:

1. Use of taurine agent within 1 month prior to the first dose of study treatment and throughout the study;
2. Patients with positive HER-2；
3. Patients with gastrointestinal obstruction or active bleeding in the gastrointestinal tract, as well as perforation and dysphagia;
4. Patients with severe heart, lung, liver, kidney, endocrine, hematopoietic system or psychiatric diseases were considered not suitable for the study group;
5. Human immunodeficiency virus (HIV) infection or known acquired immune deficiency syndrome (AIDS) or autoimmune disease or immunosuppressant use；
6. There are patients who may increase the risk of participating in the study and study medication, or other severe, acute and chronic diseases, and are not suitable for participating in the clinical study according to the judgment of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | Through study completion, Within 1 week after operation
  To evaluate the pathologic complete response rate of locally advanced gastric cancer treated with concurrent serplulimab with chemotherapy with or without taurine supplementation.

SECONDARY OUTCOMES:
R0 resection rate | Through study completion, Within 1 week after operation
  The surgical margin is microscopically-negative for residual tumor.
Major pathological response (MPR) | Through study completion, Within 1 week after operation
  Residual tumor cells below 10% in the resected specimen.
Objective response rate (ORR) | Through study completion, an average of 1 year.
  ORR is defined as the proportion of subjects with complete response (CR) or partial response (PR) according to RECIST 1.1 criteria.
Disease-free survival (DFS) | Through study completion, an average of 1 year
  DFS was defined as the time from surgery to postoperative recurrence or death from any cause, whichever occurred first. DFS was censored on the last tumor assessment date for patients still alive and without recurrence.
Event-free survival (EFS) | Through study completion, an average of 1 year
  EFS was the time from enrollment to recurrence or death from any cause. EFS was censored on the last tumor assessment date for patients still alive and without recurrence.
Overall survival (OS) | Through study completion, an average of 1 year
  OS was the time from enrolment to death from any cause. OS was censored on the last date known to be alive for patients without documentation of death.
Quality of life | Through study completion, an average of 1 year]
  The quality of life was assessed by European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30, EORTC QLQ-STO22 and Piper Fatigue Scale.
Changes in CD8+ T cell infiltration in tumor tissue | 1 year
  Changes in number, effector (TNF-α, IFN-γ, etc.) production and immune checkpoint molecule (PD-1, CTLA-4, etc.) expression of tumor-infiltrating CD8+ T cells in gastric cancer endoscopic biopsy or surgical resection material assessed via flow cytometry and immunohistochemistry.
Changes in CD8+ T cell death and function | Through study completion, an average of 1 year
  Changes in number, apoptosis rate, effector (TNF-α, IFN-γ, etc.) production and immune checkpoint molecule (PD-1, CTLA-4, etc.) expression of CD8+ T cells in peripheral venous blood assessed via flow cytometry.
Safety endpoints | Through study completion, an average of 1 year
  Number of study subjects experiencing adverse events (AEs), dose-limiting toxicities, and serious adverse events (SAEs). Safety profile will be assessed through laboratory evaluations, vital signs, and physical examinations.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Wang, MD, PhD, Study Director — Tang-Du Hospital; Xiaodi Zhao, MD, PhD, Principal Investigator — Xi-Jing Hospital; Yuanyuan Lu, MD, PhD, Principal Investigator — Xi-Jing Hospital
Locations (6):
- China (6):
  - Xi-jing Hospital, Xi'an, Shaanxi
  - Tang-Du Hospital, Xi'an, Shaanxi
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Xi 'an International Medical Center Hospital, Xi'an, Shaanxi
  - The Second Affilated Hospital Of Xi'an Jiaotong University (Xibei Hospital), Xi'an, Shaanxi
  - Xi'an NO.3 hospital, Xi'an, Shaanxi